CLINICAL TRIAL: NCT04758819
Title: Comprehensive Chromosomal Testing of Trophectoderm Biopsies of Blastocysts to Improve Live Birth Rates After in Vitro Fertilization: a Prospective Randomized Trial
Brief Title: Efficiency of Comprehensive Chromosomal Testing of Trophectoderm Biopsies of Blastocysts in In Vitro Fertilization
Acronym: Devit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP 200006
Record Dates: First submitted 2020-11-30; First posted 2021-02-17 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Infertility
Keywords: embryo aneuploidy; Intracytoplasmic Sperm Injection; in vitro fertilization; Next-Generation Sequencing; randomized controlled trial
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Embryo selection according to Day 5/6 usual morphological criteria (Istanbul consensus)
- Comprehensive chromosomal Testing of Trophectoderm biopsies of Blastocysts: CTTEB group (Experimental): Trophectoderm cells will be analyzed by NGS. Culture media will also be stored for further non-invasive chromosomal testing. Embryo selection will be done according to international guidelines (www.pgdis.org; Newsletter May 27, 2019).
  Interventions: Procedure: Comprehensive chromosomal Testing of Trophectoderm biopsies of Blastocysts (CTTEB)

INTERVENTIONS:
Procedure: Comprehensive chromosomal Testing of Trophectoderm biopsies of Blastocysts (CTTEB) — In vitro Fertilization by ICSI then embryo culture until Day 5/6; all blastocysts with morphological scores compatible with TE biopsy and vitrification will be submitted to Comprehensive chromosomal Testing of Trophectoderm biopsies of Blastocysts (CTTEB) and vitrified.
  Arms: Comprehensive chromosomal Testing of Trophectoderm biopsies of Blastocysts: CTTEB group

SUMMARY:
Preimplantation embryo aneuploidy is a major source of adverse outcomes in human reproduction since it leads to implantation failure, early pregnancy loss or severe chromosomal diseases. The risk of embryos aneuploidy is drastically increased after 35 years old. The intra uterine transfer of euploid embryos assessed through such techniques as next-generation sequencing (NGS) based Comprehensive chromosomal Testing of Trophectoderm (TE) biopsies of Blastocysts (CTTEB), may improve implantation and live birth rates, and decrease miscarriage rates. But no randomized controlled trial (RCT) was ever performed to test the interest of CTTEB for women that really needed it (≥35 to ≤ 41 years old). In this multicentre randomized-controlled-trial, the investigators will compare live birth rate obtained after the first single frozen-thawed blastocyst transfer cycle following the freeze-all-Intracytoplasmic sperm injection cycle in infertile and old couples between two different strategies of Day 5/6 blastocyst selection:

* Control group: morphological criteria (Istanbul consensus)
* Interventional group: international recommendations after CTTEB (www.pgdis.org; Newsletter May 27, 2019).

DETAILED DESCRIPTION:
The presence of chromosomal abnormalities (aneuploidy) in the pre-implantation embryonic stage is one of the major causes of human reproductive disorders, as it is responsible for embryo implantation failures, early or late miscarriages and the birth of children with chromosomal syndromes. This is mainly due to the existence of chromosomal abnormalities of meiotic, especially maternal, or mitotic origin occurring during the first three cell divisions of the embryo. As a result, human embryos have higher rates of aneuploidy than other species. Thus, it has been suggested that only 30% of conceptions reach term.

The objective of Assisted Reproductive Technologies (ART) is to optimize the chances of conception and delivery of healthy new-borns. It is necessary to improve the results of IVF (in vitro fertilization) programs and to reduce adverse effects (miscarriages, multiple pregnancies), especially in couples with patients with poor prognosis, such as older women. The choice of embryos to be transferred is a key step for the success of ART infertility treatments.

Currently, the choice of embryos is based solely on their morphology, evaluated on the 5th or 6th day of development at a stage known as the "blastocyst". Each embryo is observed under the microscope and described according to standardized morphological criteria. This description of the blastocyst is based on 3 constituents of the embryo: the degree of expansion of the blastocoelic cavity, the appearance of the internal cell mass (ICM) and the presence of trophectodermal cells (TE). These criteria have been described as predictive of live birth rates after transfer of fresh or thawed embryos. However, its ability to identify the embryo with the highest potential for implantation is debatable, due to its weak association with embryonic chromosomal status, which is a critical factor in the implant potential of each embryo. In addition, it is known that embryos that do not meet these morphological criteria are discarded, although it has been proven that their transfer could lead to a live birth.

Since the risk of embryonic aneuploidy is significantly increased after the age of 35, the objective of our RCT is to evaluate the efficacy of the CTTEB using the latest technologies and methodologies (i.e., combined embryo culture to blastocyst stage, immediate freezing of the embryonic cohort with delayed transfer, TE biopsy, NGS, and Single Embryo Transfer (SET)) in the management of infertile patients over 35 years of age. The live birth rate obtained after the first transfer of a single frozen embryo will be compared between two groups of couples, randomized in two arms: i) transfer of a single euploid blastocyst; ii) transfer of a single blastocyst of unknown chromosomal status, chosen on the basis of the usual morphological criteria, in the first thawing cycle following the freezing of all the blastocysts of the patient couples.

In addition, the culture medium of each embryo collected will be analysed in a second stage to assess whether it is possible to develop a diagnosis of aneuploidy without the need for trophectoderm biopsy (non invasive).

ELIGIBILITY:
Inclusion Criteria

Women :

* Age ≥35 to ≤ 41 years old (according to date of birth at time of informed consent) who are eligible for ovarian stimulation and ART treatment, including intracytoplasmic sperm injection (ICSI)
* BMI=18-35 kg/m2 inclusive
* No intrauterine and/or endometrial abnormalities that would interfere with implantation or pregnancy (for instance polyp, fibroid, …)

Inclusion Criteria Men:

* Use of ejaculated motile sperm (donated and/or cryopreserved sperm is allowed)
* Age ≤ 50 years old

Inclusion Criteria Couples:

* Primary or secondary infertility
* Dated and signed inform consent
* Affiliated to National Insurance
* French speaking, able to understand the study

Criteria after randomization

Couple having at least one blastocyst with morphological score on Day 5/6 of in vitro embryo development (blastocoel expansion ≥3 and inner cell mass graded A, B or C and trophectoderm graded A or B

Exclusion Criteria:

Women:

* Recurrent implantation failure (previous transfer of least 5 good grade blastocysts in at least 3 fresh or frozen cycles)
* Personal history of recurrent miscarriages (more than two miscarriages)
* Altered ovarian reserve: Identified risk of poor ovarian response (history of oocyte puncture with less than 3 oocytes) or AMH<1.1 ng/mL and AFC<5)
* Presence of non isolated uni- or bilateral hydrosalpinx
* History or presence of ovarian, uterine or mammary cancer
* Contraindication to being pregnant and/or carrying a pregnancy to term
* Women with uterine polyps diagnosed during COS
* Known allergy or hypersensitivity to human gonadotropin preparations or to compounds that are structurally similar to any of the other medications administered during the trial
* Substance abuse that would interfere with trial conduct, as determined by the investigator
* Pregnant patient, nursing patient

Men:

- Use of testicular or epididymal sperm

Couples:

* Known infection with human immunodeficiency virus, active hepatitis B or C virus in the female or male partner
* Scheduled for an embryo transfer on day 2 or 3
* Embryo freezing refusal
* Scheduled for a fresh embryo transfer
* Scheduled with an egg donation
* Scheduled with autologous oocytes thawing
* Scheduled for a preimplantation genetic diagnosis
* Participation in another ART clinical trial within the past 30 days
* Participation with another interventional study involving human subjects

Exlusion criteria to check on randomization day :

- Women with less than 3 follicles ≥ 14 mm on the triggering day or the day before the triggering

Ages: 35 Years to 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of live birth | One year
  To compare live birth rate (LBR) obtained after the first single frozen-thawed blastocyst transfer cycle following the freeze-all-Intracytoplasmic sperm injection (ICSI) cycle

SECONDARY OUTCOMES:
Number of live birth taking in consideration further single frozen-thawed blastocyst cycles | Until 48 months
  To compare live birth rate between both groups from the time where couples are randomized, i.e. in intention to treat principle, taking in consideration further single frozen-thawed blastocyst cycles during the studied period ("cumulative live birth" rate limited to the studied period)
Biological ICSI parameters | 30 months (inclusion period)
  Biological ICSI parameters will be assessed using a composite variable defined by:
  * Number of oocyte retrievals without blastocyst and/or blastocysts vitrification
  * Number of cryopreserved Day 5 and/or Day 6 blastocysts
  * Number of blastocysts still cryopreserved at the end of the study
Pregnancy outcome | 18 months (participation period)
  Pregnancy parameters will be assessed using a composite variable defined by:
  - Implantation rate (ratio between gestational sacs and transferred embryo)
  * Rate of started (hCG>100UI/ml) per oocyte retrieval
  * Rate of started (hCG>100UI/ml) per embryo transfer
  * Rate of clinical pregnancy (defined by at least one gestational sac at ultrasound) per oocyte retrieval
  * Rate of clinical pregnancy (defined by at least one gestational sac at ultrasound) per embryo transfer
  * Rate of ongoing (≥ 12 WA) pregnancy per oocyte retrieval
  * Rate of ongoing (≥ 12 WA) pregnancy per embryo transfer
Ratio between the proportion of women with live birth and days after randomization | Until 48 months
  - Ratio between the proportion of women with live birth and days after randomization
Cost of the procedure | 18 months (participation period)
  To compare cost of the procedure between both groups and estimate a cost per additional live birth
Efficiency of non-invasive chromosomal testing | Until 48 months
  Direct cost of non-invasive chromosomal testing, in blastocyst culture conditioned medium, as compared to the referent standard one, after TE biopsies and total cost .
obstetrical parameters | 18 months (participation period)
  obstetrical parameters will be assessed using a composite variable defined by:
  * Miscarriage, defined as a clinical pregnancy loss that occurs before 20 WA;
  * Pre-eclampsia, defined as gestational hypertension (Blood pressure ≥ 14 mm Hg systolic or ≥ 9 mm Hg diastolic,associated with proteinuria ≥ 0.3 grams (300 mg) or more of protein in a 24-hour urine sample
Perinatal parameters: | 18 months (participation period)
  Perinatal parameters defined by:
  * gestational age (in WA)
Perinatal parameters: | 18 months (participation period)
  Perinatal parameters defined by:
  • biometry (weight (g))
Perinatal parameters: | 18 months (participation period)
  Perinatal parameters defined by:
  * height (cm)
  * head circumference (cm) according to the sex of newborns
Perinatal parameters: | 18 months (participation period)
  Perinatal parameters defined by:
  • Apgar score at 1 and 5mn after birth (/10)
Perinatal parameters: | 18 months (participation period)
  Perinatal parameters defined by:
  * Number or children admitted in admission to neonatal intensive care unit
Perinatal parameters: | 18 months (participation period)
  Perinatal parameters defined by:
  • Number of children with major malformations defined according to the European register EUROCAT)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Frydman, Pharm D, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (10):
- France (10):
  - Hôpital Jean Verdier, Bondy
  - Hôpital Antoine Béclère, Clamart
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Cochin, Paris
  - Hopital Tenon, Paris
  - CHU Strasbourg, Schiltigheim
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No